CLINICAL TRIAL: NCT00006508
Title: Disorders of Systemic Glucose Balance
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Center for Research Resources (NCRR) (NIH)
Purpose: Diagnostic
Other Study IDs: NCRR-M01RR00036-0770; M01RR000036 (NIH)
Record Dates: First submitted 2000-11-18; First posted 2000-11-20 (Estimated); Last update posted 2005-06-24 (Estimated); Status verified 2003-12

CONDITIONS: Hypoglycemia
MeSH Terms: conditions — Hypoglycemia

INTERVENTIONS:
Procedure: Controlled hypoglycemia using insulin
Procedure: formula meal

SUMMARY:
We wish to identify people with hypoglycemia (low blood sugar) and ultimately determine why the blood sugar levels are so low. To do so, we will contrast the responses of patients suspected to have hypoglycemia with those of healthy subjects during standardized tests. Those tests may include: 1) a controlled hypoglycemia produced by administration of insulin, a blood sugar-lowering hormone, and sugar, 2) a formula meal, and 3) a period of up to 72 hours without food.

ELIGIBILITY:
Inclusion Criteria:

* Patients with suspected hypoglycemia
* Healthy subjects (controls)
* Absence of known macrovascular disease or of known CNS disease by medical history, physical examination or ECG (exclusions for induced hypoglycemia)
* Ability to give informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult

CONTACTS AND LOCATIONS:
Locations (1):
- Washington University, St Louis, Missouri, United States